CLINICAL TRIAL: NCT05055011
Title: Parental Attitudes and Beliefs Regarding Risks Associated With Opioid Use in Children
Brief Title: Parental Attitudes and Beliefs Regarding Risks Associated With Opioid Use in Children With Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-1169; NCI-2021-01159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1169 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-01; First posted 2021-09-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey, medical record review): Parents complete survey over 20 minutes. Patients' medical records are reviewed.
  Interventions: Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Review of medical records
Other: Survey Administration — Complete survey

SUMMARY:
This study investigates parents' attitudes and beliefs on the risks of opioid use in children with cancer. Pain is the common symptom reported by pediatric cancer patients. Opioids are the mainstay in the treatment of cancer-related pain. Despite an almost universal desire to prevent or mitigate pain in their children, parents exhibit complex behaviors from withholding prescribed opioids entirely to giving less than the prescribed analgesic dose of opioid to discontinuing despite ongoing pain. Information gathered from this study may help address a crucial knowledge gap in researchers' understanding of parental attitudes and beliefs regarding the risks associated with opioid use in children and adolescents.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine parents' level of concern regarding the use of opioids for pain in their children.

SECONDARY OBJECTIVES:

I. To explore differences in parents' level of concern regarding the use of opioids for pain in their children as well as level of concern for side effect of opioids between the opioid subgroup and non-opioid subgroup.

II. To explore differences in other parental attitudes and beliefs between the opioid subgroup and the non-opioid subgroup.

III. For each concern, associations between:

IIIa. Level of concern regarding the use of opioids and the age and disease of the child.

IIIb. Level of concern regarding the use of opioids and parental history of addiction.

IIIc. Level of concern regarding the use of opioids and a family history of addiction.

OUTLINE:

Parents complete survey over 20 minutes. Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Parents must be at least 18 years old
* The parent must be able to understand, read, write, and speak English
* The parent must provide verbal informed consent
* The child of the parents must be 18 years old or younger
* The child must have a diagnosis of cancer

Exclusion Criteria:

A non-cancer diagnosis (neurofibromatosis, Li-Fraumeni syndrome for example).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents whose children are on or have been on an opioid for cancer-related pain and parents whose children have not been on an opioid for cancer-related pain
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Parents' level of concern regarding the use of opioids for pain in their children. | through study completion, an average of 1 year
  Will be summarized using proportion along with a 95% confidence interval in opioid subgroup and non-opioid subgroup separately.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Madden, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org